CLINICAL TRIAL: NCT02063256
Title: 7 NUTS Study . A Randomized Dietary Intervention Trial on the Influence of Diet on Human Sperm Quality in Subfertile Men.
Brief Title: 7 NUTS Study. Diet Modification and Male Fertility.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Aldo Maina, MD Internal Medicine Obstetric Medicine, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS93-2013
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Male Subfertility; Oligospermia; Asthenospermia; Teratospermia
Keywords: sperm count; sperm concentration; mobility; diet; PUFA (polyunsaturated fatty acids)
MeSH Terms: conditions — Infertility, Male; Oligospermia; Asthenozoospermia; Teratozoospermia | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7 NUTS a day (Active Comparator): the patients allocated to this arm will be instructed to supplement their diet with 7 nuts a day (whole shelled weight around 75 grams)
  Interventions: Dietary Supplement: 7 nuts a day
- Diet modification (Experimental): the patients allocated to this arm will be instructed to modify their diet allowing more intake of PUFA rich food avoiding saturated fat rich food
  Interventions: Other: Diet modification

INTERVENTIONS:
Dietary Supplement: 7 nuts a day — add 7 nuts a day (whole shelled weight 75 grams) to standard diet
  Arms: 7 NUTS a day
Other: Diet modification — modify the diet allowing more intake of PUFA rich food and cutting the consumption of saturated fatty acids
  Arms: Diet modification

SUMMARY:
Setting. Outpatient fertility clinic.

Aim. Investigate if a modification in nutritional habits may improve in the short term the qualities of human sperm, testing two hypothesis:

i) that adding to the diet a natural whole food rich in polyunsaturated fatty acids (PUFA)

OR

ii) that reducing the intake of saturated fatty acids and increasing the consumption of PUFA may affect beneficially sperm parameters.

Population. N. 100 hypofertile male subjects attending a fertility clinic.

Type of study. Interventional study. No drugs or pharmacologic supplementation will be required nor allowed.

Two different type of intervention are scheduled:

* Supplementation to western style diet with nuts, naturally rich in PUFA
* Diet modification increasing intake of PUFA-rich foods and cutting the consumption of food rich in saturated fats.

Protocol

* Baseline visit and recruiting.
* Informed consent
* Randomized allocation to treatment group in a 1: 1 manner

Blinding. Investigators deputed to sperm analysis and statistician are blinded as to type of intervention.

Phases:

* i) basal
* ii) after 15 weeks That interval is chosen because encompasses an entire spermatogenesis cycle.

Outcomes. Primary

* sperm count, concentration,morphology and mobility.

Secondary:

* serum folate assay,
* plasma PUFA (ALA, EPA, DHA) assay,
* body weight and BMI variation

Statistics. A comparison for all sperm parameters (count,concentration,morphologic abnormalities, mobility) will be carried out by an analysis within groups and within patient.

DETAILED DESCRIPTION:
The planned trial is nutritional based only, with a modification of diet in order to obtain an increase of PUFA intake with/without a reduction of saturated fatty acid intake.

Two different types of intervention are scheduled:

* Supplementation to western style diet with food naturally rich in PUFA
* Diet modification, increasing intake of PUFA naturally rich foods and cutting the consumption of saturated fats.

The supplementation is obtained adding 7 nuts a day to regular diet. The diet modification is obtained by increasing intake of nuts and seeds (walnuts, hazelnuts, almonds, peanuts, sesame, sunflower, flaxseed) and derived oils, fish and vegetables; cutting the consumption of processed meat and dairy products is required as well.

The type of diet or supplementation is supported by oral and written information. The compliance to diet will be followed by administration of validated questionnaires.

The effect of the diet modifications will be followed by a number of plasma biomarkers we plan to compare at baseline and post intervention. The body weight and BMI will be checked, as both types of intervention are intended to not affect significantly mean body weight.

ELIGIBILITY:
Inclusion Criteria:

* sperm concentration > 5.000.000 ml
* progressive motile forms < 35%
* BMI < 30
* normal FSH (Follicle Stimulating Hormone reference values 1-10 IU)

Exclusion Criteria:

* allergy to nuts or seeds
* clinical varicocele
* recent surgery for varicocele
* vasectomy

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
sperm count | 15 weeks
  Change in sperm count from baseline to 15 weeks
sperm concentration | 15 weeks
  change in sperm concentration from baseline to 15 weeks
sperm motility | 15 weeks
  change in sperm motility (% of progressive forms) from baseline to 15 weeks
sperm morphology | 15 weeks
  change in sperm morphology ( % normal forms ) from baseline to 15 weeks

SECONDARY OUTCOMES:
change in weight (BMI) | 15 weeks
  change in body weight (BMI) from baseline to 15 weeks
Change in serum cholesterol | 15 weeks
  change in serum cholesterol levels from baseline to 15 weeks
change in serum folate | 15 weeks
  change in serum folate from baseline to 15 weeks
change in plasma alpha linolenic acid (ALA) levels | 15 weeks
  change in ALA levels from baseline to 15 weeks
change in plasma eicosapentaenoic acid (EPA) | 15 weeks
  change in plasma EPA levels from baseline to 15 weeks
change in plasma docosahexaenoic acid (DHA) | 15 weeks
  change in plasma DHA levels from baseline to 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Maina, MD, Principal Investigator — Ospedale Sant'Anna Medicina Interna. Azienda Ospedaliera Universitaria Città della Salute e della Scienza Torino Italy
Locations (1):
- Ospedale Sant'Anna. Dipartimento di Ostetricia e Neonatologia. S.C. Biochimica Clinica "Baldi e Riberi" Settore Malattie Metaboliche - Dipartimento di Medicina di Laboratorio A.O.U. Citta' della Salute e della Scienza Presidio San Giovanni Battista - Moli, Torino, Italy